CLINICAL TRIAL: NCT04112056
Title: Post-market Surveillance Study of an Infant Formula Containing Moderately Hydrolyzed Protein and Low Lactose: A Before-after Trial
Brief Title: Post-market Surveillance Study of an Infant Formula Containing Moderately Hydrolyzed Protein and Low Lactose
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Collaborators: Huantai Maternal and Child Health Care Hospital (Unknown)
Responsible Party: Principal Investigator, Jianmeng Liu, Professor in Perinatal Epidemiology, Peking University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PKUFM.191010
Record Dates: First submitted 2019-09-26; First posted 2019-10-02 (Actual); Last update posted 2020-04-02 (Actual); Status verified 2020-03

CONDITIONS: Infant Nutrition Disorders; Gastrointestinal Dysfunction
Keywords: Mild gastrointestinal disorders; Infant formula; Infant gastrointestinal symptoms questionnaire
MeSH Terms: conditions — Infant Nutrition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study formula (Experimental): The infants recruited are provided with the study formula named NAN Comfort producted by Nestle Deutschland AG, Werk Biessenhofen containing moderately hydrolyzed protein and low lactose for free during study, and asked to drink the study formula more than half of the total diet daily.
  Interventions: Dietary Supplement: Drink the study formula (NAN Comfort producted by Nestle Deutschland AG)

INTERVENTIONS:
Dietary Supplement: Drink the study formula (NAN Comfort producted by Nestle Deutschland AG) — It is same as that stated in arm description.

SUMMARY:
The study is a before-after trial to evaluate whether the study formula containing moderately hydrolyzed protein and low lactose will be able to improve mild gastrointestinal disorders (MGDs) in infants. The study plans to recruit 90 infants between 7 days and 6 months old in Huantai Maternal and Child Health Care Hospital in Shandong Province and intervene for 14 consecutive days. On Day 0 (the time of enrolling group, but the intervention which infants recruited are asked to drink study formula begins on Day 1), Day 7, Day 14, Infant Gastrointestinal Symptoms Questionnaire-13 (IGSQ-13) is used to collect infants gastrointestinal comfort, related behaviors and other information.

DETAILED DESCRIPTION:
Mild gastrointestinal disorders in infants belong to the category of functional gastrointestinal disorders. It refers that the infants fed with formula have mild digestive dysfunction that can not be explained by organic lesions or biochemical abnormalities, mainly including intestinal colic, spitting milk, diarrhea, constipation, etc. Mild gastrointestinal disorders are common in infants aged 0 to 1 year old. A study across 15 cities in China on the prevalence of common gastrointestinal disorders in infants shows that about 1/3 of the infants have one or more types of gastrointestinal disorders, among of which diarrhea and spitting milk are most common, and most of them occur within the age of 6 months. To solve this problem, a special kind of formulas for infants containing moderately hydrolyzed protein and low lactose has been developed, and our study formula is one of them. The study formula has been already marketed in China and passed the test hosted by the comprehensive testing center of the Chinese academy of inspection and quarantine, but whether it can significantly improve the mild gastrointestinal disorders in Chinese infants remains to be evaluated.

The purpose of the study is to evaluate whether the study formula containing moderately hydrolyzed protein and low lactose will be able to improve mild gastrointestinal disorders (MGDs) in infants. After informed consent, 90 infants between 7 days and 6 months old with mild gastrointestinal disorders are included and asked to drink the study formula for 14 consecutive days as intervention. On Day 0 (the time of enrolling group, but the intervention begins on Day 1), Day 7, Day 14, the information on gastrointestinal comfort and related behaviors is collected through the Infant Gastrointestinal Symptoms Questionnaire-13 (IGSQ-13). Information on feeding, family background, anthropometric measurements and defecation is also collected. The primary endpoint of this study is gastrointestinal comfort calculated by IGSQ-13. The secondary endpoints include crying frequency, spitting milk frequency, flatulence frequency, stool frequency and consistency score, formula acceptability and satisfaction, adverse event, etc.

ELIGIBILITY:
Inclusion Criteria:

* Obtaining the informed consent of infants' parents or guardians
* Term infants (≥37 gestational weeks)
* Healthy infants aged 7-180 days
* Formula feeding or mixed feeding
* With mild gastrointestinal disorders
* Drinking the study formula more than half of the total diet daily

Exclusion Criteria:

* Adding new auxiliary food in the latest week
* Any kind of probiotics is being used
* Using drugs
* Using the formula being studied
* Having a history of milk protein allergies according to parents' reports
* Can not follow the research plans

Ages: 7 Days to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2019-10-10 (Actual); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-05-15 (Estimated)

PRIMARY OUTCOMES:
Infant Gastrointestinal Symptoms Questionnaire-13 (IGSQ-13) Index Score | On Day 0 (the time of enrolling group)
  The IGSQ-13 is a validated instrument (Riley, Trabulsi et al. 2015) consisting of 5 GI symptoms and GI-related behavioural domains. Parents (caregivers) are asked to recall specific symptoms experienced in the past week. Possible index scores range from 13 to 65; higher scores indicate higher GI burden, while lower scores indicate less GI burden.
Infant Gastrointestinal Symptoms Questionnaire-13 (IGSQ-13) Index Score | On Day 7
  The IGSQ-13 is a validated instrument (Riley, Trabulsi et al. 2015) consisting of 5 GI symptoms and GI-related behavioural domains. Parents (caregivers) are asked to recall specific symptoms experienced in the past week. Possible index scores range from 13 to 65; higher scores indicate higher GI burden, while lower scores indicate less GI burden.
Infant Gastrointestinal Symptoms Questionnaire-13 (IGSQ-13) Index Score | On Day 14
  The IGSQ-13 is a validated instrument (Riley, Trabulsi et al. 2015) consisting of 5 GI symptoms and GI-related behavioural domains. Parents (caregivers) are asked to recall specific symptoms experienced in the past week. Possible index scores range from 13 to 65; higher scores indicate higher GI burden, while lower scores indicate less GI burden.

SECONDARY OUTCOMES:
Crying frequency | On Day 0, Day 7 and Day 14
  Collected by Infant Gastrointestinal Symptoms Questionnaire-13 (IGSQ-13)
Spitting milk frequency | On Day 0, Day 7 and Day 14
  Collected by Infant Gastrointestinal Symptoms Questionnaire-13 (IGSQ-13)
Flatulence frequency | On Day 0, Day 7 and Day 14
  Collected by Infant Gastrointestinal Symptoms Questionnaire-13 (IGSQ-13)
Stool frequency and consistency | On Day 1, Day 2 and Day 3
  Collecting infants stool photos
Formula acceptability and satisfaction | On Day 14
  Collected by a structured questionnaire，which is designed for this study specially, including 5 questions, and will be analyzed separately for each question (no total score used).
Adverse event frequency | Day1 to Day 14
  Confirmed by doctor

CONTACTS AND LOCATIONS:
Overall Officials: Jian-meng Liu, PhD, Study Chair — Peking University; Ying-chao Mu, BD, Study Director — Huantai Maternal and Child Health Care Hospital
Locations (1):
- Huantai Maternal and Child Health Care Hospital, Zibo, Shandong, China

REFERENCES:
- [Derived] Huang Y, Zhou Y, Li H, Chen Y, Mu Y, Yuan A, Yang Y, Liu J. The Effects of a Partially Hydrolyzed Formula with Low Lactose and Probiotics on Mild Gastrointestinal Disorders of Infants: A Single-Armed Clinical Trial. Nutrients. 2021 Sep 25;13(10):3371. doi: 10.3390/nu13103371. PMID 34684372